CLINICAL TRIAL: NCT02646254
Title: MYOCARDIAL PROTECTION AND CLINICAL OUTCOME IN PATIENTS UNDERGOING TETRALOGY OF FALLOT REPAIR: A RANDOMIZED STUDY OF TWO CARDIOPLEGIC TECHNIQUES
Brief Title: Myocardial Protection and Clinical Outcome in Patients Undergoing Tetralogy of Fallot Repair : A Randomized Study of Two Different Cardioplegia Technique
Acronym: TOF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SUNDER LAL NEGI (Unknown)
Responsible Party: Sponsor-Investigator, SUNDER LAL NEGI, Fellow, Cardiac anesthesia., Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NK/1840/DM/16940
Record Dates: First submitted 2015-12-24; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Myocardial Protection in TOF Repair
Keywords: tetralogy of fallot, cardioplegia
MeSH Terms: conditions — Tetralogy of Fallot | interventions — Del Nido cardioplegia solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- blood cardioplegia (Active Comparator): these patients received blood cardioplegia
  Interventions: Other: blood cardioplegia
- del nido cardioplegia (Active Comparator): these patients received del nido cardioplegia
  Interventions: Other: del nido cardioplegia

INTERVENTIONS:
Other: blood cardioplegia
  Arms: blood cardioplegia
Other: del nido cardioplegia
  Arms: del nido cardioplegia

SUMMARY:
Myocardial protection and clinical outcome in patients Undergoing tetralogy of fallot repair: a randomized study of Two cardioplegic techniques.

DETAILED DESCRIPTION:
Del Nido cardioplegia has not been used for myocardial protection and clinical outcome in patients undergoing tetralogy of Fallot repair, so the investigators hypothesized that a del Nido cardioplegia technique may be beneficial in the pediatric patients undergoing tetralogy of fallot repair.

ELIGIBILITY:
Inclusion Criteria:

* Tetralogy of fallot

Exclusion Criteria:

* TOF with absent pulmonary valve , TOF with pulmonary atresia

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
inotropic score | First 24 hours
Creatine kinase MB level baseline preoperative and postoperative 0, 6, 24, and 72 hours | 72hrs
resumption of spontaneous rhythm after aortic cross clamp off | 10 minutes

SECONDARY OUTCOMES:
duration of mechanical ventilation in hours | 48 hours
ICU stay | 7 days
hospital mortality | 30 days
echocardiographic assessment | 6 months